CLINICAL TRIAL: NCT05364853
Title: Neurodevelopmental Effects of Antiseizure Medications (NEAM) - UG3 Phase
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not receive funding.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kimford Jay Meador, Professor of Neurology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 65669
Record Dates: First submitted 2022-04-21; First posted 2022-05-06 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Testing (Other): In this arm, participants will undergo the neuropsychological assessment of interest (DAYC-2) in-person.
  Interventions: Behavioral: In-Person Testing
- Remote Testing (Other): In this arm, participants will undergo the neuropsychological assessment of interest (DAYC-2) remotely over video/telehealth.
  Interventions: Behavioral: Remote Testing

INTERVENTIONS:
Behavioral: In-Person Testing — Participants will be randomly assigned to have either in-person testing of the DAYC-2 conducted. They will then cross over into the other testing condition approximately 3 weeks after their first assessment.
  Arms: In-Person Testing
Behavioral: Remote Testing — Participants will be randomly assigned to have either remote testing of the DAYC-2 conducted. They will then cross over into the other testing condition approximately 3 weeks after their first assessment.
  Arms: Remote Testing

SUMMARY:
To compare in-person to remote video assessments in children to determine the reliability of remote evaluations for future neuropsychological assessments and set a precedent for future investigations.

ELIGIBILITY:
Inclusion Criteria:

1. Parents able to provide informed consent for themselves and their child
2. Access to computer and reliable internet connection for remote testing
3. Child of women with epilepsy who was taking antiseizure medications during the pregnancy of the child being enrolled into the current study
4. Child between the ages of 24 months and 30 months of age
5. Primary language is English

Exclusion Criteria:

1. Child unable to complete the cognitive assessment (e.g., expected IQ<70)
2. Child with a major medical condition (e.g., epilepsy, diabetes, heart disease, active cancer)
3. Child who use centrally active medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Developmental Assessment of Young Children-2nd edition (DAYC-2) Standard Scores of the Communication Domain as a Measure of Direct Comparison of the 2 Testing Conditions. | Change from the first, baseline assessment to the second assessment, 21 days later.
  Standardized Scores of DAYC-2 Communication Domain at end of each period for each intervention (i.e., in-person testing and remote testing). The standard score indicates the deviation away from a reference population. A standard score of 100 is equal to the mean. Numbers less than 100 indicate poor cognitive performance compared to the mean and numbers greater than 100 represent higher cognitive performance compared to the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Kimford J Meador, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: Undecided